CLINICAL TRIAL: NCT04421235
Title: Growing Together: Expanding Knowledge About and Evaluating Services for Incarcerated Pregnant and Postpartum Women in Arkansas
Brief Title: Expanding Knowledge About and Evaluating Services for Incarcerated Pregnant and Postpartum Women in Arkansas
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 260265; UL1TR003107 (NIH)
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Health Problems in Pregnancy; Childbirth Problems; Maternal Care Patterns; Quality of Life; Emotional Stress; Health Care Acceptability; Health Risk Behaviors; Parent-Child Relations
Keywords: Incarcerated Women; Prison
MeSH Terms: conditions — Stress, Psychological; Patient Acceptance of Health Care; Health Risk Behaviors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Childbirth Support: Women who enroll in the intervention portion of this study will receive the childbirth support elements for which they are eligible in and elect to participate. Possible program elements include prenatal education classes, support group, lactation program, doula support, and parenting classes.
  Interventions: Behavioral: Childbirth support

INTERVENTIONS:
Behavioral: Childbirth support — There are 5 program components that women may receive as a part of childbirth support:
  Prenatal education - consists of up to 8 sessions of education on pregnancy, childbirth, and postpartum health and wellness.
  Support group - semi-structured group which provides time for women to process their pregnancy and postpartum-related experiences with other women facing similar challenges. Integrates mindfulness exercises, cognitive-behavioral skills, and special topics as requested by group members.
  Lactation program - program for women who wish to provide breastmilk for infants from which they are separated.
  Doula support program - 2 prenatal and 2 postnatal individual visits with a doula who will also provide continuous childbirth support and support during separation from infants.
  Parenting classes - group classes focused on helping women learn parenting skills and (if applicable) meet state requirements for reunification with children

SUMMARY:
The number of women who are incarcerated in the U.S. has increased dramatically over the past 20 years-over 750%, or from 13,258 in 1980 to 111,616 in 2016. Arkansas incarcerates 92 women per 100,000 population compared to 57 per 100,000 average across all states, ranking the state as the 8th highest in the nation. Over 75% of incarcerated women are of childbearing age and about 4% are pregnant upon intake. However, little is known about the population of women who have become incarcerated while pregnant in Arkansas - including the outcomes of these women and their children and how these outcomes may vary in relation to services that are received during incarceration. This research study aims to first expand knowledge on incarcerated women in Arkansas by using administrative data to retrospectively examine the health status and outcomes of pregnant women who were incarcerated in state prison by Arkansas from June 1, 2014 to May 31, 2019 (a five-year cohort; Aim 1). Then, we will lay the groundwork for and subsequently analyze data on outcomes and perspectives of women who have been incarcerated in Arkansas while pregnant (Aims 2 and 3). We will also seek to understand the feasibility and acceptability of elements of an enhanced support program for incarcerated pregnant women recently launched via a collaboration between Arkansas Department of Corrections and UAMS.

ELIGIBILITY:
Inclusion Criteria:

* Women incarcerated in Arkansas state prison system
* 18 years or older
* Able to give informed consent
* Pregnant or has given birth in past year

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of administrative data on women who were: 1) incarcerated in the Hawkins Unit at Wrightsville Prison between June 1, 2014 to May 31, 2019 (a five-year cohort prior to initiation of Growing Together) and 2) who received pre- and/or post-natal health care services during that incarceration.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Program Utilization | Up to 12 months after delivery
  % of eligible women who choose to enroll in each program component
Program Acceptability | Up to 12 months after delivery
  Self-report ratings of the acceptability of each program component

SECONDARY OUTCOMES:
Depressive Symptoms | Up to 12 months after delivery
  Self-report scores on Patient Health Questionnaire (PHQ-9)
Depressive Symptoms | Up to 12 months after delivery
  Self-report scores on the Edinburgh Postnatal Depression Scale
PTSD Symptoms | Up to 12 months after delivery
  Self-report scores on PTSD Checklist (PCL-5)
Drug Use | Up to 12 months after delivery
  Binary self-report for common classes of drugs
Health-Related Quality of Life | Up to 12 months after delivery
  Self-report scores on Quality of Life Scale (QOLS)
Health-Related Quality of Life | Up to 12 months after delivery
  Self-report scores on the EQ-5D-5L
Social Support | Up to 12 months after delivery
  Self-report scores on Multidimensional Scale of Perceived Social Support
Parental Stress | Up to 12 months after delivery
  Self-report scores on the Parenting Stress Index
Parental Sense of Competence | Up to 12 months after delivery
  Self-report scores on the Parenting Sense of Competence Scale
Pregnancy Complications | From the date of enrollment until the date of childbirth or the date of pregnancy loss or termination, whichever came first, assessed up to 50 weeks
  Chart review to determine presence/absence of common pregnancy complications
Childbirth Complications | Up to 12 months after delivery
  Chart review to determine presence/absence of common pregnancy complications

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Zielinski, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No